CLINICAL TRIAL: NCT02256137
Title: A Longitudinal Assessment of Frailty in Young Adult Survivors of Childhood Cancer
Status: Active, not recruiting | Type: Observational
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: FRAILTY; R01CA174851 (NIH)
Record Dates: First submitted 2014-10-01; First posted 2014-10-03 (Estimated); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Acute Lymphoblastic Leukemia; Brain Tumor; Hodgkin Lymphoma
Keywords: Frailty phenotype; Physical fitness; Childhood cancer; Late onset of chronic health conditions; Physical frailty
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Brain Neoplasms; Hodgkin Disease; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Childhood Cancer Survivors: This study will evaluate 1493 members of the St. Jude Lifetime Cohort Study (SJLIFE) who have completed a baseline functional assessment six or less years ago when 18-45 years of age.

SUMMARY:
Advances in cancer therapies have led to increasing numbers of adult survivors of pediatric malignancy. Unfortunately, treatment of childhood cancer continues to require agents designed to destroy malignant cell lines, and normal tissue is not always spared. While early treatment- related organ specific toxicities are not always apparent, many childhood cancer survivors report symptoms that interfere with daily life, including exercise induced shortness of breath, fatigue and reduced capacity to participate in physical activity. These symptoms may be a hallmark of premature aging, or frailty. Frailty is a phenotype most commonly described in older adults; it indicates persons who are highly vulnerable to adverse health outcomes. Frailty may help explain why nearly two thirds of childhood cancer survivors have at least one severe chronic health condition 30 years from diagnosis, why childhood cancer survivors are more likely than peers to be hospitalized for non-obstetrical reasons, and why they have mortality rates more than eight times higher than age-and-gender matched members of the general population.

Frailty is a valuable construct because it can be distinguished from disability and co-morbidity, and is designed to capture pre-clinical states of physiologic vulnerability that identify individuals most at risk for adverse health outcomes. These investigators have recently presented data indicating that impaired fitness is present in survivors of childhood acute lymphoblastic leukemia, brain tumor and Hodgkin lymphoma. This is relevant because frailty, characterized by a cluster of five measurements of physical fitness, is predictive of chronic disease onset, frequent hospitalization, and eventually mortality in both the elderly and in persons with chronic conditions. Using a frailty phenotype as an early predictor of later chronic disease onset will allow identification of childhood and adolescent cancer survivors at greatest risk for adverse health. An early indicator of those at risk for adverse health will allow researchers to test, and clinicians to provide, specific interventions designed to remediate functional loss, and prevent or delay onset of chronic health conditions. The investigators goals include characterizing physical frailty over a five year time span in a population of young adult survivors of childhood cancer, as well as assessing the association between frailty and the increase in the number and severity of chronic health conditions.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

* Evaluate the change in the proportion of young adult cancer survivors who are frail from baseline to a point five years later.
* Evaluate the association between frailty and worsening of chronic health conditions.
* Describe the association between demographic and treatment factors and risk for prevalent frailty.
* Estimate the effects of physical activity, diet and smoking on risk for prevalent frailty.

Participants will complete a study questionnaire to assess social support, complete body composition studies, walking speed test, physical activity monitoring, and difficulties in daily activities due to health condition. In addition, any data collected as part of the SJLIFE protocol, including questionnaires, medical history and physical, height and weight measurements, physical functioning assessment results (i.e. hand grip strength), and neuropsychological evaluation results, may also be used as part of the evaluation for this study. The information collected for this study will be compared to information collected at a previous SJLIFE clinic visit within the previous 6 years.

ELIGIBILITY:
Inclusion Criteria:

* Enrollment on the SJLIFE protocol.
* Completed baseline assessment between July 1, 2008 and June 30, 2015.
* Completed the baseline assessment between the ages of 18-45.

Exclusion Criteria:

* Currently pregnant (assessed by serum pregnancy test).
* Currently receiving treatment for cancer.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: This study will evaluate 1493 members of the St. Jude Lifetime Cohort Study (SJLIFE) who have completed a baseline functional assessment six or less years ago when 18-45 years of age.
Sampling Method: Non-Probability Sample
Enrollment: 1564 (Actual)
Dates: Start 2014-10-08 (Actual); Primary Completion 2018-09-21 (Actual); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Change in proportion of participants who are frail from baseline to 5 years later | Baseline and 5 years later (± 1 year)
  We will use McNemar's test to assess if the prevalence of frailty has significantly increased over the 5-year time period.
Association between frailty at baseline and worsening of chronic health conditions 5 years later | Baseline and 5 years later (± 1 year)
  The event of interest, worsening of chronic condition, will be defined as binary outcome which will take value of 1 if, compared to baseline evaluation, a survivor develops a new chronic condition (grade ≥3) or if the chronic condition worsens over the 5-year time period (i.e. goes from grades 1-2 to grade ≥3 or dies due to chronic condition); otherwise it will take a value of 0.
Association between demographic and treatment factors and lifestyle on prevalent frailty. | 5 years (± 1 year) after baseline evaluation
  We will examine the association in a path model (all variables are measured) as lifestyle factors are likely to be mediators of the association between treatment and the frailty outcome at the five year time point. Sex, age at diagnosis, radiation exposure, specific chemotherapy agent doses, and age will be included in the initial theoretical model as exogenous variables and physical activity, diet, smoking status and frailty will be included as endogenous variables. Other variables, like medication use, baseline chronic disease, etc. will be evaluated for their contributions to the outcomes.
Effects of physical activity, diet and smoking on prevalent frailty | 5 years (± 1 year) after baseline evaluation
  We will examine the association in a path model (all variables are measured) as lifestyle factors are likely to be mediators of the association between treatment and the frailty outcome at the five year time point. Sex, age at diagnosis, radiation exposure, specific chemotherapy agent doses, and age will be included in the initial theoretical model as exogenous variables and physical activity, diet, smoking status and frailty will be included as endogenous variables. Other variables, like medication use, baseline chronic disease, etc. will be evaluated for their contributions to the outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Kirsten Ness, PT, PhD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols